CLINICAL TRIAL: NCT05514054
Title: EMBER-4: A Randomized, Open-Label, Phase 3 Study of Adjuvant Imlunestrant vs Standard Adjuvant Endocrine Therapy in Patients Who Have Previously Received 2 to 5 Years of Adjuvant Endocrine Therapy for ER+, HER2- Early Breast Cancer With an Increased Risk of Recurrence
Brief Title: A Study of Imlunestrant Versus Standard Endocrine Therapy in Participants With Early Breast Cancer
Acronym: EMBER-4
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18459; J2J-MC-JZLH (Other: Eli Lilly and Company); 2022-501007-28 (EudraCT Number)
Record Dates: First submitted 2022-08-23; First posted 2022-08-24 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Imlunestrant; Tamoxifen; Anastrozole; Letrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Imlunestrant (Experimental): Imlunestrant administered orally.
  Interventions: Drug: Imlunestrant
- Investigator's Choice of Endocrine Therapy (Active Comparator): Investigator's choice of tamoxifen, anastrozole, letrozole, or exemestane administered per local approved label.
  Interventions: Drug: Tamoxifen; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane

INTERVENTIONS:
Drug: Imlunestrant — Administered orally.
  Other Names: LY3484356
  Arms: Imlunestrant
Drug: Tamoxifen — Administered per local approved label.
  Arms: Investigator's Choice of Endocrine Therapy
Drug: Anastrozole — Administered per local approved label.
  Arms: Investigator's Choice of Endocrine Therapy
Drug: Letrozole — Administered per local approved label.
  Arms: Investigator's Choice of Endocrine Therapy
Drug: Exemestane — Administered per local approved label.
  Arms: Investigator's Choice of Endocrine Therapy

SUMMARY:
The main purpose of this study is to measure how well imlunestrant works compared to standard hormone therapy in participants with early breast cancer that is estrogen receptor positive (ER+) and human epidermal receptor 2 negative (HER2-). Participants must have already taken endocrine therapy for two to five years and must have a higher-than-average risk for their cancer to return. Study participation could last up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of ER+, HER2- early-stage, resected, invasive breast cancer without evidence of distant metastasis.
* Participants must have received at least 24 months but not more than 60 months of any adjuvant ET, from time of adjuvant ET initiation.
* Participants may have received (neo) adjuvant chemotherapy and/or targeted therapy with a CDK4/6- or PARP- inhibitor.
* Must have an increased risk of disease recurrence based on clinical-pathological risk features.
* Have a Performance Status of 0 or 1 on the Eastern Cooperative Oncology Group scale.
* Have adequate organ function.

Exclusion Criteria:

* Have any evidence of metastatic disease (including contralateral ALN) or inflammatory breast cancer at primary breast cancer diagnosis.
* Participants with more than a 6-month consecutive gap in therapy during the course of prior adjuvant ET.
* Participants who have completed or discontinued prior adjuvant ET >6 months prior to screening.
* Participants with a history of previous breast cancer are excluded, with the exception of ipsilateral DCIS treated by locoregional therapy alone ≥5 years ago.
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 180 days after the last dose of study intervention.
* Participant has previously received ET of any duration for breast cancer prevention (tamoxifen or AIs) or raloxifene.
* Participants with a history of any other cancer.
* Have serious preexisting medical conditions that, in the judgment of the investigator, would preclude participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-Free Survival (IDFS) | Randomization to recurrence or death from any cause (up to 10 years)
  IDFS excluding second non-breast primary invasive cancers

SECONDARY OUTCOMES:
Distant Recurrence-Free Survival (DRFS) | Randomization to Distant Recurrence or Death from Any Cause (up to 10 Years)
  DRFS
Overall Survival (OS) | Randomization to Death from Any Cause (up to 10 Years)
  OS
Pharmacokinetics (PK): Steady State Plasma Concentrations of Imlunestrant | Year 1, Month 2 to Month 4
  PK: steady state plasma concentrations of imlunestrant
Change from Baseline in the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core Questionnaire (EORTC QLQ-C30) Physical Functioning | Visit 1 Day 1 up to end of Year 5
  The EORTC QLQ-C30 is a 30-question patient reported instrument used to assess multidimensional quality of life (QOL) in cancer patients. It consists of 15 domains: 1 global QOL scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). Physical functioning was measured by items 1 to 5. The sum score was linearly transformed to the range 0 - 100 as recommended by the EORTC (higher score is better).
Change from Baseline in the EORTC QLQ-C30 Role Functioning | Visit 1 Day 1 up to end of Year 5
  The EORTC QLQ-C30 is a 30-question patient reported instrument used to assess the multidimensional QOL in cancer patients. It consists of 15 domains: 1 global QOL scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). Role functioning was measured by items 6 and 7. The sum score was linearly transformed to the range 0 - 100 as recommended by the EORTC (higher score is better).
Change from Baseline in the EORTC QLQ-C30 Global QOL | Visit 1 Day 1 up to end of Year 5
  The EORTC QLQ-C30 is a 30-question patient reported instrument used to assess the multidimensional QOL in cancer patients. It consists of 15 domains: 1 global QOL scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). Global QOL was measured by items 29 and 30. The sum score was linearly transformed to the range 0 - 100 as recommended by the EORTC (higher score is better).
Proportion of Time on Study Treatment with High Overall Adverse Event Burden | Visit 1 Day 1 up to end of Year 5
  FACT GP5 = Functional Assessment of Cancer Therapy - General Physical Well-being Item 5 (FACT GP5). High overall adverse event burden is defined as a score of 3 or 4 on a 5-point Likert scale. Higher scores represent higher symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (671):
- United States (136):
  - USO - Southern Cancer Center, Daphne, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - Infirmary Cancer Care, Mobile, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - USO - Arizona Oncology Associates - HAL, Glendale, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic in Arizona - Phoenix, Phoenix, Arizona
  - TMC HealthCare, Tucson, Arizona
  - The University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - UCSF - John Muir Health Cancer Center Berkeley, Berkeley, California
  - Washington Health, Fremont, California
  - Chao Family Comprehensive Cancer Center and Ambulatory Care (CIACC) - Irvine, Irvine, California
  - Loma Linda University Cancer Center, Loma Linda, California
  - Pacific Cancer Care, Monterey, California
  - St. Joseph Hospital, Orange, California
  - University of California, Irvine (UCI) Health - UC Irvine Medical Center, Orange, California
  - University of California Davis (UC Davis) Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente San Diego Mission Road, San Diego, California
  - Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - Saint Joseph's Medical Center, Stockton, California
  - Anschutz Cancer Pavilion, Aurora, Colorado
  - UCHealth Memorial Hospital, Colorado Springs, Colorado
  - UCHealth Harmony, Fort Collins, Colorado
  - Banner MD Anderson Cancer Center at North Colorado Medical Center, Greeley, Colorado
  - USO - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Banner MD Anderson Cancer Center at McKee Medical Center, Loveland, Colorado
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - AdventHealth Altamonte Springs, Altamonte Springs, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Millennium Oncology Research Clinic, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - USO - Cancer Care Centers of Brevard, Palm Bay, Florida
  - USO - Woodlands Medical Specialists, Pensacola, Florida
  - Miami Cancer Institute - Plantation, Plantation, Florida
  - Tampa General Hospital, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Summit Cancer Care, PC, Savannah, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Simmons Cancer Institute at SIU, Springfield, Illinois
  - The University of Kansas Cancer Center - Westwood, Westwood, Kansas
  - Ochsner Clinic Foundation, Covington, Louisiana
  - Pontchartrain Cancer Center, Hammond, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - York Hospital, York Village, Maine
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - Southcoast Centers for Cancer Care, Fairhaven, Massachusetts
  - Dana-Farber Cancer Institute - Foxborough, Foxborough, Massachusetts
  - Dana-Farber Cancer Institute - Merrimack Valley, Methuen, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional Medical Center, Milford, Massachusetts
  - Mass General Cancer Center at Newton-Wellesley, Newton, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center - South Shore Hospital, South Weymouth, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - M Health Fairview Cancer Clinic -Edina, Edina, Minnesota
  - USO - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Allina Health Cancer Institute, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Minnesota, Rochester, Minnesota
  - University of Missouri Hospital, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Dana-Farber - New Hampshire Oncology/Hematology, Londonderry, New Hampshire
  - MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - Astera Cancer Care, East Brunswick, New Jersey
  - Regional Cancer Care Associates, Little Silver, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Capital Health Medical Center - Hopewell, Pennington, New Jersey
  - New Mexico Oncology Hematology Consultants Ltd., Albuquerque, New Mexico
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - New York Oncology Hematology Associate, Albany, New York
  - Maimonides Cancer Center, Brooklyn, New York
  - NYU Langone Health - Brooklyn, Brooklyn, New York
  - R.J. Zuckerberg Cancer Center, Lake Success, New York
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island, Mineola, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Laura and Isaac Perlmutter Cancer Center, New York, New York
  - NYC Health + Hospitals / Bellevue, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Queens Medical Associates, Queens, New York
  - University of Rochester - Wilmot Cancer Institute, Rochester, New York
  - Phelps Hospital, Sleepy Hollow, New York
  - Staten Island University Hospital, Staten Island, New York
  - Clinical Research Alliance, Westbury, New York
  - Messino Cancer Center, Asheville, North Carolina
  - Aultman Hospital, Canton, Ohio
  - USO - Oncology Hematology Care, Cincinnati, Ohio
  - Mercy Health - St. Vincent Medical Center, Toledo, Ohio
  - Good Samaritan Regional Medical Center, Corvallis, Oregon
  - USO - Oncology Associates of Oregon, Eugene, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - USO - Compass Oncology, Tigard, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - USO - Alliance Cancer Specialists, PC, Horsham, Pennsylvania
  - Thomas Jefferson University - Clinical Research Institute, Philadelphia, Pennsylvania
  - Lifespan Cancer Institute, Providence, Rhode Island
  - St Francis Cancer Center, Greenville, South Carolina
  - The West Clinic, PLLC dba West Cancer Center, Germantown, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - USO - Texas Oncology, Austin, Texas
  - USO - Texas Oncology, Dallas, Texas
  - USO - Texas Oncology, Denison, Texas
  - Texas Oncology - West Texas, El Paso, Texas
  - William Beaumont Army Medical Center, El Paso, Texas
  - USO - Texas Oncology, Flower Mound, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - John Peter Smith Hospital, Fort Worth, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - USO - Texas Oncology, Fort Worth, Texas
  - USO - Texas Oncology, Fredericksburg, Texas
  - USO - Texas Oncology, McAllen, Texas
  - USO - Texas Oncology, Plano, Texas
  - Scott & White Hospital - Round Rock, Round Rock, Texas
  - Mays Cancer Center, San Antonio, Texas
  - Baylor Scott & White Medical Center - Temple, Temple, Texas
  - US Oncology Research Network, The Woodlands, Texas
  - USO - Texas Oncology, Webster, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia
  - Bon Secours St. Francis Medical Center, Midlothian, Virginia
  - USO - Virginia Oncology Associates, Norfolk, Virginia
  - USO - Virginia Cancer Specialists, Reston, Virginia
  - USO - Oncology & Hematology Associates of Southwest Virginia, Roanoke, Virginia
- Argentina (20):
  - Centro de Oncología e Investigación de Buenos Aires, Berazategui
  - Centro de Investigaciones Medicas y Desarrollo LC, Buenos Aires
  - Investigaciones Clinicas Moleculares (ICM), Buenos Aires
  - Centro Oncologico Korben, Buenos Aires
  - CIPREC, Buenos Aires
  - Mautalen Salud e Investigación, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Instituto Alexander Fleming, Buenos Aires
  - Clinica Adventista Belgrano, CABA
  - Centro Medico Privado CEMAIC, Capital
  - Fundación CORI para la Investigación y Prevención del Cáncer, La Rioja
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata
  - Fundacion Scherbovsky, Mendoza
  - Instituto Médico Río Cuarto, Río Cuarto
  - Fundacion Estudios Clinicos, Rosario
  - Centro Polivalente de Asistencia e Investigacion Clinica - CER San Juan, San Juan
  - Instituto San Marcos, San Juan
  - Exelsus Oncología Clínica, San Miguel de Tucumán
  - Go Centro Medico San Nicolás, San Nicolás
  - Clinica Viedma S. A, Viedma
- Australia (22):
  - Ballarat Health Services, Ballarat Central
  - Box Hill Hospital, Box Hill
  - Monash Health, Clayton
  - Coffs Harbour Health Campus, Coffs Harbour
  - St Vincent's Hospital, Darlinghurst
  - Barwon Health, Geelong
  - Royal Hobart Hospital, Hobart
  - Launceston General Hospital, Launceston
  - Liverpool Hospital, Liverpool
  - Mackay Base Hospital, Mackay
  - St Vincent's Hospital, Melbourne
  - Northern Hospital, Melbourne
  - Maroondah Hospital, Melbourne
  - Breast Cancer Research Centre-WA, Nedlands
  - Lake Macquarie Private Hospital, Newcastle
  - Goulburn Valley Health, Shepparton
  - Gold Coast University Hospital, Southport
  - Mater Hospital Sydney, Sydney
  - Royal Darwin Hospital, Tiwi
  - The Townsville Hospital, Townsville
  - Hervey Bay Hospital, Urraween
  - The Queen Elizabeth Hospital, Woodville
- Austria (6):
  - Medizinische Universität Graz, Graz
  - Uniklinikum Salzburg, Salzburg
  - Private Practice - Dr. Hubalek, Schwaz
  - Medizinische Universität Wien, Vienna
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
  - Klinik Hietzing, Vienna
- Belgium (17):
  - Institut Jules Bordet, Anderlecht
  - CHIREC - site delta, Auderghem
  - CHU Saint-Pierre, Brussels
  - Centre Hospitalier Universitaire Brugmann, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - Jessa Ziekenhuis, Hasselt
  - Jan Yperman Ziekenhuis, Ieper
  - AZ Groeninge Campus Kennedylaan, Kortrijk
  - Groupe Jolimont, La Louvière
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman, Liège
  - CHU UCL Namur/Site Sainte Elisabeth, Namur
  - AZ Oostende vzw, Ostend
  - Clinique Saint Pierre, Ottignies
  - AZ Nikolaas, Sint-Niklaas
  - CHR Verviers - La Tourelle, Verviers
- Brazil (36):
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos
  - CTO - Centro de Tratamento Oncológico, Belém
  - Oncocentro de Minas Gerais, Belo Horizonte
  - Hospital Sirio Libanes, Brasília
  - Centro Integrado de Oncologia de Curitiba, Curitiba
  - Centro de Pesquisa Clínica do Instituto do Câncer do Ceará, Fortaleza
  - Hospital Araújo Jorge, Goiânia
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia, Ijuí
  - Hospital de Cancer de Londrina, Londrina
  - Hospital Moinhos de Vento, Porto Alegre
  - Centro Gaucho Integrado De Oncologia, Hematologia, Ensino E Pesquisa, Porto Alegre
  - Hospital São Lucas da PUCRS, Porto Alegre
  - Hospital de Amor Amazônia, Porto Velho
  - Multihemo, Recife
  - Hospital de Clínicas de Ribeirão Preto, Ribeirão Preto
  - Instituto Nacional de Câncer - INCA, Rio de Janeiro
  - Hospital São Lucas de Copacabana, Rio de Janeiro
  - Centro de Tratamento de Tumores Botafogo para Oncoclinicas Rio de Janeiro SA, Rio de Janeiro
  - Instituto de Educação, Pesquisa e Gestão em Saúde, Rio de Janeiro
  - Nucleo de Oncologia da Bahia, Salvador
  - Faculdade de Medicina do ABC, Santo André
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
  - IPITEC, São Paulo
  - NotreDame Intermedica Saude S.A, São Paulo
  - Instituto de Ensino e Pesquisa São Lucas, São Paulo
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo
  - Hospital Sírio Libanês, São Paulo
  - Clínica de Pesquisa e Centro de Estudos em Ginecologia Oncológica e Mamária LTDA, São Paulo
  - Hospital BP, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - A. C. Camargo Cancer Center, São Paulo
  - Núcleo de Pesquisa Clínica da Rede São Camilo, São Paulo
  - Instituto de Assistência Médica ao Servidor Público Estadual - IAMSPE/HSPE-FMO Conhecer Centro de Oncolog -T, São Paulo
  - Instituto D'Or de Pesquisa e Ensino (IDOR), São Paulo
  - Hospital Santa Paula, São Paulo
  - CEDOES, Vitória
- Canada (9):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary
  - Victoria Hospital & Children's Hospital - London Health Sciences Centre, London
  - Centre Hospitalier de l'Université de Montréal, Montreal
  - Jewish General Hospital, Montreal
  - Centre intégré universitaire de santé et de services sociaux du Nord-de-l'Île-de-Montréal (CIUSSS NÎM) - H -T, Montreal
  - CHU de Québec-Université Laval, Hôpital du Saint-Sacrement, Québec
  - BC Cancer Surrey, Surrey
  - Humber River Hospital, Toronto
  - Sunnybrook Research Institute, Toronto
- China (51):
  - Anyang Cancer Hospital, Anyang
  - Affiliated Hospital of Hebei University, Baoding
  - Beijing Hospital, Beijing
  - Cancer Hospital Chinese Academy of Medical Science, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Friendship Hospital Affiliate of Capital University, Beijing
  - The First Hospital of Jilin University, Changchun
  - The First People's Hospital of Changde City, Changde
  - Xiangya Hospital Central South University, Changsha
  - Hunan Cancer Hospital, Changsha
  - Sichuan Cancer hospital, Chengdu
  - Deyang City People's Hospital, Deyang
  - Dongguan People's Hospital, Dongguan
  - Shunde Hospital of Southern Medical Univesity, Foshan
  - Fujian Medical University Union Hospital-1 Bingfanglou, Fuzhou
  - The 900th Hospital of the Joint Logistics Support Force of the Chinese People's Liberation Army, Fuzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Guangdong Maternity and Child Health Care Hospital, Guangzhou
  - Hainan General Hospital, Haikou
  - The First People's Hospital of Hangzhou, Hangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - First Huai'an Hospital Affiliated to Nanjing Medical University, Huai'an
  - Huizhou Municipal Central Hospital, Huizhou
  - Jiangmen Center Hospital, Jiangmen
  - Jinan Central Hospital, Jinan
  - Jining Medical University - Affiliated Hospital, Jining
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang
  - The Third Hospital of Nanchang, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - The Second People's Hospital of Neijiang, Neijiang
  - Hwa Mei Hospital University of Chinese Academy of Sciences, Ningbo
  - Ningbo First Hospital, Ningbo
  - Fudan University Shanghai Cancer Center, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou
  - ShenZhen People's Hospital, Shenzhen
  - Shenzhen Second People's Hospital, Shenzhen
  - Cancer Hospital Chinese Academy of Medical Sciences. Shenzhen Center, Shenzhen
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University Cancer Institute & Hospital, Tianjing
  - Xinjiang Medical University Cancer Hospital - Urumqi, Ürümqi
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Hubei Cancer Hospital, Wuhan
  - Wannan Medical College Yijishan Hospital, Wuhu
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Xiangyang Central Hospital, Xiangyang
  - The Central Hospital of Yongzhou - North Campus, Yongzhou
  - The First People's Hospital of Yueyang, Yueyang
  - Yuncheng Central Hospital - Eastern Hospital, Yuncheng
  - Central Hospital of Guangdong Provincial Agricutural Reclamation, Zhanjiang
- Czechia (8):
  - Masarykuv onkologicky ustav, Brno
  - Nemocnice Horovice, Hořovice
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Ostrava, Ostrava
  - Multiscan, Pardubice
  - Fakultni Thomayerova nemocnice, Prague
  - Fakultni nemocnice Motol, Prague
  - Fakultni nemocnice Bulovka, Prague
- France (34):
  - Sainte Catherine Institut du Cancer Avignon Provence, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - CHU Besançon, Besançon
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux
  - CHRU de Brest, Brest
  - Pole Santé République, Clermont-Ferrand
  - Henri Mondor Hospital, Créteil
  - Polyclinique De Blois, La Chaussée-Saint-Victor
  - CHD Vendee, La Roche-sur-Yon
  - Groupe Hospitalier La Rochelle-Ré-Aunis - Hôpital Saint Louis, La Rochelle
  - Chu Grenoble Alpes, La Tronche
  - Clinique Victor Hugo Le Mans, Le Mans
  - Clinique Francois Chenieux, Limoges
  - Hopital Prive Jean Mermoz, Lyon
  - Centre Hospitalier Régional Metz Thionville - Hôpital de Mercy, Metz
  - Centre Hospitalier Intercommunal de Mont-de-Marsan et du Pays des Sources, Mont-de-Marsan
  - Centre de Cancérologie du Grand Montpellier, Montpellier
  - Polyclinique de Gentilly, Nancy
  - Centre Antoine-Lacassagne, Nice
  - Hôpital Saint-Louis, Paris
  - Groupe hospitalier Paris saint Joseph, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Institut Curie, Paris
  - Hôpital Tenon, Paris
  - Centre Hospitalier de Pau, Pau
  - Centre Catalan d'Oncologie, Perpignan
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Institut Jean Godinot, Reims
  - Institut Curie - site Saint-Cloud, Saint-Cloud
  - Centre Hospitalier Privé Saint-Grégoire, Saint-Grégoire
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Centre de cancérologie des Dentellières, Valenciennes
  - Institut de Cancérologie de Lorraine Alexis Vautrin, Vandœuvre-lès-Nancy
- Germany (34):
  - Gemeinschaftspraxis hop-augsburg, Augsburg
  - Universitaetsklinikum Augsburg, Augsburg
  - Praxisklinik Krebsheilkunde fur Frauen, Berlin
  - Onkologische Schwerpunktpraxis Kurfuerstendamm, Berlin
  - Helios Klinikum Berlin-Buch, Berlin
  - Marienhospital Bottrop, Bottrop
  - Universitaetsklinikum Koeln, Cologne
  - Städtisches Klinikum Dessau, Dessau
  - Onkologiezentrum Donauwörth, Donauwörth
  - St.-Johannes-Hospital Dortmund, Dortmund
  - MVZ Medical Center Düsseldorf GmbH, Düsseldorf
  - Universitaetsklinikum Erlangen, Erlangen
  - Kliniken Essen-Mitte, Evangelische Huyssens-Stiftung, Essen
  - Agaplesion Markus Krankenhaus, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Private Practice - Dr. Helmut Oettle und Prof.Dr.med. Frank Mayer, Friedrichshafen
  - SRH Wald-Klinikum Gera, Gera
  - OSP Göttingen, Göttingen
  - St. Anna Hospital, Herne
  - Universitaetsklinikum des Saarlandes, Homburg
  - Klinikverbund Allgäu gGmbH, Kempten
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Zentrum fuer ambulante gynaekologische Onkologie (ZAGO), Krefeld
  - Universitätsmedizin Mannheim, Mannheim
  - Onkologisch-hämatologisches Forschungsinstitut am Habsburgring, Mayen
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen, München
  - Klinikum Ernst von Bergmann, Potsdam
  - HELIOS Kliniken Schwerin, Schwerin
  - Robert-Bosch-Krankenhaus, Stuttgart
  - SRH Zentralklinikum Suhl, Suhl
  - Klinikum Mutterhaus der Borromäerinnen, Trier
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaetsklinikum Ulm, Ulm
  - Helios HSK Wiesbaden, Wiesbaden
- Greece (14):
  - Agios Savvas Regional Cancer Hospital, Athens
  - Alexandra Hospital, Athens
  - IASO Obstetrics - Gynecology Clinic, Athens
  - Iaso Private General Obstetrics Gynecological & Pediatric Clinic Diagnostic Therapeutic & Research Center -T, Athens
  - Attikon General University Hospital, Chaïdári
  - University General Hospital of Heraklion, Heraklion
  - University Hospital of Ioannina, Ioannina
  - University General Hospital of Larissa, Larissa
  - General Oncology Hospital of Kifissia "Agioi Anargiroi", Nea Kifissia
  - Olympion General Clinic, Pátrai
  - University Hospital of Patras, Pátrai
  - BioClinic Thessaloniki, Thessaloniki
  - Agios Loukas Clinic, Thessaloniki
  - European Interbalkan Medical Center, Thessaloniki
- Queen Mary Hospital, Hksar, Hong Kong
- Hungary (5):
  - Országos Onkológiai Intézet, Budapest
  - Uzsoki Utcai Kórház, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Bacs-Kiskun Megyei Korhaz, Kecskemét
  - Szabolcs Szatmár Bereg Vármegyei Oktatókórház, Nyíregyháza
- India (18):
  - Hemato Oncology Clinic, Ahmedabad
  - KD Hospital, Ahmedabad
  - Medstar Speciality Hospital, Bangalore
  - KLES Dr. Prabhakar Kore Hospital & M.R.C, Belagavi
  - All India Institute of Medical Sciences, Bhubaneswar
  - Postgraduate Institute of Medical Education & Research, Chandigarh
  - Cancer Institute (WIA), Chennai
  - Nizam's Institute of Medical Sciences, Hyderabad
  - Regency Hospital, Kanpur
  - Krishna Institute of Medical Sciences - Karad, Karad
  - Kolhapur Cancer Centre Private Limited, Kolhāpur
  - Tata Memorial Hospital, Mumbai
  - Rashtrasant Tukdoji Regional Cancer Hospital, Nagpur
  - Delhi State Cancer Institute, New Delhi
  - Grant Medical Foundation - Ruby Hall Clinic, Pune
  - Lifepoint Multispeciality Hospital, Pune
  - Regional Cancer Centre - Thiruvananthapuram, Thiruvananthapuram
  - Mahatma Gandhi Cancer Hospital and Research Institute, Visakhapatnam
- Ireland (9):
  - Bon Secours Cork Hospital, Cork
  - Cork University Hospital, Cork
  - St. Vincent's University Hospital, Dublin
  - St. James's Hospital, Dublin
  - UCD School of Medicine Beacon Hospital, Dublin
  - Beaumont Hospital, Dublin, Dublin
  - Galway University Hospital, Galway
  - Sligo General Hospital, Sligo
  - Waterford Regional Hospital, Waterford
- Israel (8):
  - Carmel Hospital, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
  - Yitzhak Shamir Medical Center, Ẕerifin
- Italy (20):
  - Aou Ospedali Riuniti Umberto I, Ancona
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - IRCCS - AOU di Bologna, Bologna
  - Ospedale Antonio Perrino, Brindisi
  - Istituto di Candiolo IRCCS - Fondazione del Piemonte per l'Oncologia, Candiolo
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale San Martino, Genova
  - Ospedale Generale Provinciale Macerata, Macerata
  - Istituto Europeo di Oncologia IRCCS, Milan
  - Humanitas Istituto Clinico Catanese, Misterbianco
  - Azienda Ospedaliero Universitaria, Modena
  - Ospedale San Gerardo-ASST Monza, Monza
  - University of Naples Federico II, Naples
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Istituto Nazionale Tumori Regina Elena, Rome
  - Humanitas, Rozzano
  - Ospedale San Giovanni Moscati, Statte
  - Azienda Ospedaliera Santa Maria Terni, Terni
- Japan (50):
  - Juntendo University Hospital, Bunkyō City
  - Chiba University Hospital, Chiba
  - Chiba cancer center, Chiba
  - St. Luke's International Hospital, Chūōku
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Fukushima Medical University, Fukushima
  - Fukuyama City Hospital, Fukuyama
  - Gifu University Hospital, Gifu
  - Tokai University Hachioji Hospital, Hachioji-shi
  - Kansai Medical University Hospital, Hirakata
  - Hiroshima City Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Shimane University Hospital, Izumo
  - Sagara Hospital, Kagoshima
  - Kameda Clinic, Kamogawa
  - Ishikawa Prefectural Central Hospital, Kanazawa
  - St. Marianna University Hospital, Kawasaki
  - Japanese Foundation for Cancer Research, Kōtō City
  - Kumamoto Breast Surgical Hospital, Kumamoto
  - Kumamoto Shinto General Hospital, Kumamoto
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
  - Kyoto University Hospital, Kyoto
  - Shinshu University Hospital, Matsumoto
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - Miyazaki Prefectural Miyazaki Hospital, Miyazaki
  - Kanazawa Medical University Hospital, Mukai-awagasaki
  - Nagoya University Hospital, Nagoya
  - Nagoya City University Hospital, Nagoya
  - Naha Nishi Clinic, Naha
  - Niigata Cancer Center Hospital, Niigata
  - Hyogo Medical University Hospital, Nishinomiya
  - Okayama University Hospital, Okayama
  - Nakagami Hospital Okinawa, Okinawa
  - National Hospital Organization - Osaka National Hospital - Institute For Clinical Research, Osaka
  - Gunma Prefectural Cancer Center, Otashi
  - Kitasato University Hospital, Sagamihara
  - Saitama Red Cross Hospital, Saitama
  - National Hospital Organization Hokkaido Cancer Center, Sapporo
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Showa Medical University Hospital, Shinagawa City
  - National Center for Global Health and Medicine, Shinjyuku-ku
  - Shizuoka General Hospital, Shizuoka
  - National Hospital Organization Takasaki General Medical Center, Takasaki
  - Tokushima University Hospital, Tokushima
  - Tsukuba University Hospital, Tsukuba
  - Tochigi Cancer Center, Utsunomiya
  - Iwate Medical University Hospital, Yahaba-cho, Shiwa-gun
  - Yokohama City University Medical Center, Yokohama
  - Kanagawa cancer center, Yokohama
- Mexico (18):
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, Ciudad Madero
  - CIO - Centro de Inmuno-Oncología de Occidente, Guadalajara
  - Clinica de Investigacion en Reumatologia y Obesidad S. C., Guadalajara
  - Preparaciones Oncologicas, León
  - CENEIT Oncológicos. Centro Especializado en Investigación y Tratamientos Oncológicos, Mexico City
  - Grupo Medico Camino Sc, Mexico City
  - Axis Heilsa S. de R.L. de C.V., Monterrey
  - Centro Regiomontano de Investigación, Monterrey
  - Filios Alta Medicina, Monterrey
  - Oaxaca Site Management Organization, Oaxaca City
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City
  - Unidad Médica Onco-hematológica, Puebla City
  - PanAmerican Clinical Research - Querétaro - Avenida Antea, Querétaro
  - Oncologico Potosino, S.C., San Luis Potosí City
  - Centro Medico Zambrano Hellion, San Pedro Garza García
  - Hospital Angeles, Tijuana
  - Centro Oncologico Estatal ISSEMyM ( COEI ), Toluca
- Netherlands (11):
  - Wilhelmina Ziekenhuis Assen, Assen
  - Amphia Ziekenhuis, locatie Breda Molengracht, Breda
  - Reinier de Graaf Ziekenhuis, locatie Delft, Delft
  - Deventer Ziekenhuis, Deventer
  - Albert Schweitzer Ziekenhuis, locatie Dordwijk, Dordrecht
  - Ziekenhuisgroep Twente, locatie Almelo, Hengelo
  - Spaarne Gasthuis - Hoofddorp, Hoofddorp
  - Maastricht UMC+, Maastricht
  - Haga Ziekenhuis locatie Leyweg, The Hague
  - VieCuri Medisch Centrum, locatie Venlo, Venlo
  - Zaans Medisch Centrum, Zaandam
- Poland (9):
  - Szpitale Pomorskie Sp. z o. o., Gdynia
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie, Koszalin
  - Salve Medica, Lodz
  - Opolskie Centrum Onkologii w Opolu im. prof. Tadeusza Koszarowskiego, Opole
  - FORMED2, Oświęcim
  - Mazowiecki Szpital Wojewódzki w Siedlcach, Siedlce
  - MICS Centrum Medyczne Torun, Torun
  - Luxmed Onkologia sp. z o. o., Warsaw
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie, Warsaw
- Portugal (6):
  - Hopital Garcia de Orta, Almada
  - Champalimaud Foundation, Lisbon
  - Hospital da Luz Lisboa, Lisbon
  - Centro Hospitalar Universitário Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Hospital Beatriz Ângelo, Lisbon
  - Centro Hospitalar de Vila Nova de Gaia/Espinho - Unidade I, Vila Nova de Gaia
- Romania (11):
  - C.M.D.T.A. Neomed, Brasov
  - Onco Medint Srl, Bucharest
  - Lotus-Med, Bucharest
  - SC Memorial Healthcare International SRL, Bucharest
  - Spitalul Clinic Colțea, Bucharest
  - Gral Medical Diagnostic Center, Bucharest
  - Institutul Oncologic Cluj, Cluj-Napoca
  - Centrul de Oncologie "Sfântul Nectarie", Craiova
  - Radiology Therapeutic Center, Otopeni
  - Ovidius Clinical Hospital OCH, Ovidiu
  - S C Oncocenter Oncologie Clinica S R L, Timișoara
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - Raffles Hospital, Singapore
- Slovakia (2):
  - Onkologicky Ustav sv. Alzbety, Bratislava
  - Narodny onkologicky ustav, Bratislava
- South Korea (21):
  - Dongnam Institute of Radiological and Medical Sciences, Busan
  - Soon Chun Hyang University Cheonan Hospital, Cheonan-si
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Yeungnam Univeristy Medical Center, Gyeongsan-si
  - Chonnam National University Hwasun Hospital, Hwasun-gun
  - Inha University Hospital, Incheon
  - Gachon University Gil Medical Center, Namdong-gu
  - Seoul National University Bundang Hospital, Seongnam
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan
- Spain (44):
  - CHUAC-Hospital Teresa Herrera, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Torrecárdenas, Almería
  - Hospital Infanta Cristina, Badajoz
  - Parc de Salut Mar - Hospital del Mar, Barcelona
  - Hospital Quiron Barcelona, Barcelona
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Osi Bilbao-Basurto, Bilbao
  - Hospital Universitario de Burgos, Burgos
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario Getafe, Getafe
  - Hospital Universitario San Cecilio, Granada
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida
  - Hospital San Pedro, Logroño
  - Hospital Lucus Augusti, Lugo
  - Hospital La Princesa, Madrid
  - Hospital Beata María Ana, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - H.R.U Málaga - Hospital Materno-infantil, Málaga
  - Hospital Vithas Málaga, Málaga
  - Hospital Universitari Son Espases, Palma
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitari Sant Joan de Reus, Reus
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitario de Toledo, Toledo
  - Hospital Clinico de Valencia, Valencia
  - Hospital Quirónsalud Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- Taiwan (11):
  - Changhua Christian Hospital, Changhua County
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Tzu Chi General Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Hospital - Liouying Branch, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (25):
  - Adana Medical Park Seyhan Hastanesi, Adana
  - Adana City Hospital, Adana
  - Sakarya Training and Research Hospital, Adapazarı
  - Hacettepe Universitesi, Altindağ
  - Ankara Gülhane Eitim ve Aratrma Hastanesi, Ankara
  - Ankara Etlik City Hospital, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Ankara Bilkent Şehir Hastanesi, Ankara
  - Akdeniz Universitesi Hastanesi, Antalya
  - Antalya Egitim ve Arastırma Hastanesi, Antalya
  - Uludag Universitesi, Bursa
  - Dicle Üniversitesi, Diyarbakır
  - Trakya University Medical Faculty Hospital, Edirne
  - Gaziantep Universitesi Sahinbey Arastirma ve Uygulama Hastanesi, Gaziantep
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Marmara Universitesi Pendik Egitim Arastirma Hastanesi, Istanbul, Pendik
  - Ege Universitesi Hastanesi, Izmir
  - zmir Katip Çelebi Üniversitesi Atatürk Eitim Ve Aratrma Hastanesi, Izmir
  - Izmir Medical Park Hospital, Izmir, Karsiyaka
  - Kocaeli Üniversitesi, Kocaeli
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi Eğitim ve Araştırma Hastanesi, Malatya
  - Mersin University, Mersin
  - Mugla Sitki Kocman Universitesi Egitim ve Arastirma Hastanesi, Muğla
  - Ondokuz Mayıs Universitesi, Samsun
  - Medipol Mega Universite Hastanesi, Stanbul
- United Kingdom (13):
  - Colchester General Hospital, Colchester
  - Hairmyres Hospital, East Kilbride, Glasgow
  - Western General Hospital, Edinburgh
  - Clatterbridge Cancer Centre - Liverpool, Liverpool
  - St Bartholomew's Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Mount Vernon Hospital, Northwood
  - Derriford Hospital, Plymouth
  - Panthera Biopartners - Preston, Preston
  - Royal Berkshire Hospital, Reading
  - Panthera Biopartners - Manchester, Rochdale
  - Lister Hospital, Stevenage
  - Oncology Research, Wigan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Imlunestrant Versus Standard Endocrine Therapy in Participants With Early Breast Cancer (EMBER-4) — https://trials.lilly.com/en-US/trial/356295